CLINICAL TRIAL: NCT00193921
Title: A Randomised Phase II Study of Two Regimens of Palliative Chemoradiation Therapy in the Management of Locally Advanced Non Small Cell Lung Cancer
Brief Title: Chemoradiotherapy in Patients With Localised Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Collaborators: Cancer Council Queensland (Other); Victorian Cancer Council (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TROG 03.07; PMCC Protocol No. 03/85
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Non Small Cell Lung Carcinoma
Keywords: Chemoradiotherapy; High dose; palliative radiotherapy; Quality of life
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Vinorelbine; Radiotherapy; Radiation; Gemcitabine; Capecitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Vinorelbine + cisplatin + high-dose palliative radiotherapy
  Interventions: Drug: Vinorelbine; Radiation: High dose Radiotherapy; Drug: Cisplatin
- B (Active Comparator): Gemcitabine + high-dose palliative radiotherapy
  Interventions: Drug: Gemcitabine; Radiation: High Dose Radiotherapy

INTERVENTIONS:
Drug: Vinorelbine — IV, 25mg/m2, days 1, 8, 22
  Other Names: Navelbine, Vinorelbine Ebewe
  Arms: A
Radiation: High dose Radiotherapy — External beam radiation, 40 Gy/20#/5 per week
  Other Names: Radiation
  Arms: A
Drug: Gemcitabine — 200mg (flat dose) IV days 1, 8, 15
  Other Names: Gemzar, Xeloda
  Arms: B
Drug: Cisplatin — 20mg/m2, IV, weekly
  Other Names: Cisplatin Ebewe, Cisplatin Injection
  Arms: A
Radiation: High Dose Radiotherapy — External beam radiation, 30 Gy/15#/5 per week
  Other Names: Radiation
  Arms: B

SUMMARY:
The study compares 2 different methods of combined chemotherapy and radiotherapy for the treatment of localised lung cancer in patients not suitable for surgery.

Hypothesis(es) to be tested:

1. Vinorelbine + cisplatin + high-dose palliative radiotherapy is superior to gemcitabine + high dose palliative radiotherapy in terms of efficacy in a multi-institutional setting
2. Vinorelbine + cisplatin + high-dose palliative radiotherapy is superior to gemcitabine + high dose palliative radiotherapy in terms of feasibility in a multi-institutional setting
3. Vinorelbine + cisplatin + high-dose palliative radiotherapy has a favourable toxicity profile relative to gemcitabine + high-dose palliative radiotherapy

DETAILED DESCRIPTION:
A third of patients with non-small cell lung cancer (NSCLC) present with Stage IIIA or IIIB disease, which is not amenable to curative resection. Single modality local therapy, either surgery or radiation, only cures a fraction of such patients.

Radical radiation is not feasible for all patients with unresectable Stage IIIA or IIIB non-small cell lung cancer, based upon the extent of the loco-regional disease or the medical state of the patient. Patients of good performance status receiving protracted high-dose palliative radiotherapy do obtain a survival benefit from this therapy. Studies have shown a survival advantage by adding chemotherapy to radical radiation therapy: but studies in the high-dose palliative radiotherapy setting are lacking. Two regimens of concurrent chemotherapy with high-dose palliative radiotherapy have been developed locally, with established MTDs. These 2 regimens do warrant a comparative assessment in a phase II trial, prior to a phase III trial against high dose palliative radiation alone (36Gy/12#/5).

This is a randomised phase II trial comprising of 2 arms for randomization as follows:

Arm A:External beam radiation, 40 Gy/20#/5 per week, Plus concurrent Vinorelbine, IV, 25mg/m2, days 1, 8, 22 and + Cisplatin 20mg/m2, IV, weekly

Arm B:External beam radiation, 30 Gy/15#/5 per week, Plus concurrentGemcitabine, 200mg (flat dose) IV days 1, 8, 15

An equal number of patients will be randomised to each arm. The randomisation will be carried out by the Princess Alexandra Trial Centre.

Patients will be assessed at baseline, weekly during treatment, and then at 3 weeks, 6 weeks and 12 weeks post treatment then 3 monthly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven non-small cell lung cancer.
* Planned high dose palliative radiation therapy for locoregional control. Examples include patients with:

  1. Stage I - IIIB disease with

     * disease technically unsuitable for radical therapy, or · weight loss in excess of 10%, or
     * concurrent medical illness
  2. Patients found to have a locally advanced thoracic disease suitable for radical therapy but on work up are found to have a FDG-PET only solitary metastasis.
* All potential patients, prior to registration, must be reviewed at a multidisciplinary lung oncology meeting attended by medical oncologists, radiation oncologists and radiologists.
* No prior radiotherapy or chemotherapy for non-small cell lung cancer.
* ECOG performance status 0, 1.
* Adequate hepatic, bone marrow and renal function.
* If patient is female of child bearing potential, she must not be pregnant or lactating. Males and females of reproductive potential must practise adequate contraception.
* Written informed consent.

Exclusion Criteria:

* Patient unable to receive all therapy as an outpatient.
* Significant medical conditions which in the opinion of the investigator would compromise the planned delivery of the chemotherapy and radiotherapy or which may be potentially exacerbated by these modalities.
* History of any other cancer (except non-melanoma skin cancer or carcinoma in situ of the cervix) unless in complete remission and off all therapy for that cancer for at least 5 years.
* Receiving treatment with another investigational agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2003-02; Primary Completion 2009-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Objective response rate (RECIST criteria) | Final analysis will occur when all have a minimum 1 year follow-up after randomisation. Approx 3 years after start of trial.
Symptomatic response rate | Final analysis will occur when all have a minimum 1 year follow-up after randomisation. Approx 3 years after start of trial.
The feasibility (i.e. % of patients who cannot complete the planned RT dose or who require a break for toxicity) and problems encountered with protocol compliance in the setting of a multi-institutional TROG study. | Final analysis will occur when all have a minimum 1 year follow-up after randomisation. Approx 3 years after start of trial.
Toxicity of both treatments | Final analysis will occur when all have a minimum 1 year follow-up after randomisation. Approx 3 years after start of trial.

SECONDARY OUTCOMES:
Progression-free survival | Final analysis will occur when all have a minimum 1 year follow-up after randomisation. Approx 3 years after start of trial.
QOL as assessed by FACT-L version 4. | Final analysis will occur when all have a minimum 1 year follow-up after randomisation. Approx 3 years after start of trial.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Michael, Study Chair — Peter MacCallum Cancer Centre, Australia; Bryan Burmeister, Study Chair — Princess Alexandra Hospital
Locations (8):
- Australia (8):
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Mater Misericordiae Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - North Queensland Oncology Service, Townsville, Queensland
  - The John Flynn Hospital, Tugun, Queensland
  - Frankston Hospital, Frankston, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Border Medical Oncology, Wondonga, Victoria

REFERENCES:
- See also: Click here for more information about this study on the TROG official website — http://www.trog.com.au